CLINICAL TRIAL: NCT06358768
Title: Post-Partum Hemorrhage and Improvement in Technical Skills on Different Rules Using Actors Scenario
Brief Title: Post-Partum Haemorrhage (PPH) Improvement of Skills With Actor Simulations
Acronym: PPH
Status: Not yet recruiting | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Collaborators: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Claudio Celentano, Haed of unit, G. d'Annunzio University
Other Study IDs: ObGynEASC005
Record Dates: First submitted 2024-03-17; First posted 2024-04-11 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: PPH - Postpartum Hemorrhage
Keywords: PPH; actor scenario; improve skills; improve teamwork reactions
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Gynecologists: ObGyn specialists
  Interventions: Other: teamwork job improvement overall; Other: teamwork job improvement in actor scenario vs mannequin scenario
- Midwives: Midwives registered
  Interventions: Other: teamwork job improvement overall; Other: teamwork job improvement in actor scenario vs mannequin scenario
- Anesthesiologists: Anesthesiologists specialists
  Interventions: Other: teamwork job improvement overall; Other: teamwork job improvement in actor scenario vs mannequin scenario
- Surgical theatre nurse: nurse
  Interventions: Other: teamwork job improvement overall; Other: teamwork job improvement in actor scenario vs mannequin scenario
- Sanitary support personnel: SSP regularly working in labour ward
  Interventions: Other: teamwork job improvement overall; Other: teamwork job improvement in actor scenario vs mannequin scenario

INTERVENTIONS:
Other: teamwork job improvement overall — increase of teamwork capacities and skills improvement
  Other Names: skills improvement
Other: teamwork job improvement in actor scenario vs mannequin scenario — increase of teamwork capacities and skills improvement. Comparison within different roles and different scenario learning

SUMMARY:
Pre test and post test questionnaire for evaluation of skills and teamwork capacities in PPH management

DETAILED DESCRIPTION:
Obstetricians, midwives, anesthesiologists, surgical theatre nurses, and sanitary collaborators are enrolled voluntary in a teamwork (2 gynecologists, 2 midwives, 1 anesthesiologist, 1 surgical theatre nurse, and 1 sanitary collaborator) for managing a PPH scenario. 2 different teamworks will attend a frontal lecture of 30' and afterwards they attend a scenario with actors/facilitators (enrolled within ObGyn residents) or attend a scenario with a high-fidelity mannequin after a questionnaire indicating previous experiences and skills (at the end they accept video recording of the scenario and the use of data for scientific reasons). The teamwork is recorded and an extensive debriefing is conducted using the video records and a dataset indicating positive and negative approach. After they will answer a questionnaire indicating the use of this scenario and indicating how it is compared to reality. Personal approach to teamwork job is also described.

ELIGIBILITY:
Inclusion Criteria:

* personnel working in labour ward and surgical theatre
* Volunteers

Exclusion Criteria:

* none

Ages: 19 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: persons working in our hospitals
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
teamwork | 1 month
  Scoring the teamwork efficacy (1-10)
skills | 1 month
  improvement score (1-10)

SECONDARY OUTCOMES:
scenario quality | 1 month
  is the scenario adherent to reality with a score(1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Celentano, MD, Study Chair — University d'annunzio; Luisa Patanè, MD, Principal Investigator — Ospedale Giovanni XXIII Bergamo
Locations (2):
- Italy (2):
  - Claudio Celentano, Pescara, PE
  - Ospedale Giovanni XXIII, Bergamo

IPD SHARING:
Plan to Share IPD: No
not jet decided